CLINICAL TRIAL: NCT06445582
Title: Synaptic Vesicle Glycoprotein 2A-PET/CT and PET/MRI Combined Clinical Criteria Score in the Diagnosis of Early Cognitive Alteration
Brief Title: SV2A-PET/CT and PET/MRI Combined Clinical Criteria Score in the Diagnosis of Early Cognitive Alteration
Status: Not yet recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023_ky_390
Record Dates: First submitted 2024-05-22; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease
Keywords: Molecular Imaging；; Positron Emission Tomography Computed Tomography；; SV2A protein, human
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CANDI: China Aging and Neurodegenerative Initiative
  Interventions: Diagnostic Test: [18F]SDM-8

INTERVENTIONS:
Diagnostic Test: [18F]SDM-8 — synaptic vesicle glycoprotein 2 A（SV2A）PET tracer [18F]SDM-8

SUMMARY:
Using SV2A-PET to character a cohort of patients with early cognitive impairment using the novel synaptic probe 18F-labeled difluoro-analog of UCB-J（also known as 18F-SDM-8）

DETAILED DESCRIPTION:
A community-based population (Han Chinese) in Hefei, China, based on the CANDI cohort；Single-center prospective case-control study；The projected enrollment population is 80; 40 patients with Alzheimer's Disease（AD）, 30 patients with Mild Cognitive Impairment（MCI）; 10 healthy controls. Diagnostic experiments and predictive prognostic experiments with new probes.

ELIGIBILITY:
Inclusion Criteria:

* AD Group
* All diagnostic criteria for AD patients met the National Institute of Neurological Speech-Language Disorders Stroke Institute and Alzheimer's Disease and Related Disorders Association criteria;
* Comply with the American Psychiatric Association Diagnostic and Statistical Workbook of Mental Disorders, 5th edition (DSMIV);
* All subjects were unconscious and could be accompanied by behavioral and psychiatric abnormalities. Subjects who meet the above criteria are eligible for enrollment.
* Those who understand the process of this clinical trial and sign the informed consent form (in addition, non-AD volunteers will be recruited through verbal dissemination and posting of paper advertisements to serve as the non-AD control group, and the final control group will be screened by the clinician and consist of healthy people of similar age and gender).
* MCI Group
* Concerns about cognitive changes, and concerns about finding changes in comparison with one's prior level may originate from the patient himself or herself, from an informed person, or from an experienced specialist;
* Impairment of one or more cognitive areas, primarily memory, executive function, attention, language, and visuospatial function;
* Maintaining independence in daily living, there can be minor impairment in complex instrumental daily abilities;
* Absence of dementia, mild disease, and no evidence of serious impairment of social or occupational abilities;
* Presence of one of the Aβ class biomarkers and/ neuronal damage class markers detected by imaging, cerebrospinal fluid;
* All subjects and their guardians give informed consent to the study and sign the informed consent form;

Exclusion Criteria:

* With confirmed cerebrovascular disease, the presence of multiple or extensive cerebral infarcts;
* Other types of dementia: Parkinson's disease dementia, vascular dementia, frontotemporal lobe dementia, dementia with Lewy bodies;
* Sudden onset or stroke-like episodes;
* Early onset of focal neurological symptoms, such as hemiparesis, computational deficits, ataxia, or sensory loss;
* Seizures or gait abnormalities early in the onset of the disease;
* Evidence of drug applications that cause significant effects on cognitive function;
* Those who are allergic to alcohol;
* Persons with alcohol allergy; (ix) Persons with left-handedness; (x) Persons with left-handedness;
* Those with claustrophobia or other reasons for not being able to cooperate with the examination;
* Those with serious heart, liver, lung, kidney and other organ diseases, meeting the above conditions were excluded from the group.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a single-center prospective exploratory clinical trial, and given this, it is proposed to initially enroll only 80 evaluable subjects (including 40 patients with ALZHEIMER'S DISEASE, 30 patients with MILD COGNITIVE DISABILITY, and 10 age-sex matched non-ALZHEIMER 'S DISEASE controls), each subject underwent 18F-SDM-8 PET/CT imaging, the ability of the tracer to bind to SV2A in the brain as well as non-specific binding, and correlation analysis with changes in relevant clinical indicators to assess the safety and diagnostic efficacy of the tracer.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
SUVR（Standardized Uptake Value Ratio） | 1year
  Standardized semi-quantitative values of SUVR for each brain region of the cerebral cortex；Standardized Uptake Value ratio (SUVr) is a metric used to evaluate the results of PET scans of the brain. It is a measure of the extent of abnormal metabolism or abnormal deposits in a brain region by comparing the uptake value of a specific brain region to the uptake values of neighboring regions.
  SUVr is calculated as follows:
  1. first, a reference region is selected, usually an adjacent region of healthy tissue that is unaffected by disease.
  2. then, the uptake value for the region of interest (e.g., the brain region), denoted as SUV, is calculated.
  3. next, the average uptake value of the reference region, denoted as SUVref, is calculated.
  4. finally, the SUVr is calculated, obtained by dividing the SUV of the region of interest by the SUVref of the reference region.

SECONDARY OUTCOMES:
AUC（Area under the curve）of SUVR | 1year
  AUC is defined as the area under the ROC curve enclosed with the axes. ROC (receiver operating characteristic curve) receiver operating characteristic curve, is invented by electronic engineers and radar engineers in World War II used to detect enemy carriers (aircraft, ships) on the battlefield indicators, belongs to the signal detection theory.
  The SV2A SUVR calculation was performed using the reference brain region method described above, and the AUC was used to measure the ability of the SUVR to classify the AD disease spectrum versus healthy controls, and its correlation with clinical scale scores was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xie, PhD, Principal Investigator — University of Sience and Technology of China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stockburger C, Miano D, Baeumlisberger M, Pallas T, Arrey TN, Karas M, Friedland K, Muller WE. A Mitochondrial Role of SV2a Protein in Aging and Alzheimer's Disease: Studies with Levetiracetam. J Alzheimers Dis. 2016;50(1):201-15. doi: 10.3233/JAD-150687. PMID 26639968
- [Background] Bajjalieh SM, Frantz GD, Weimann JM, McConnell SK, Scheller RH. Differential expression of synaptic vesicle protein 2 (SV2) isoforms. J Neurosci. 1994 Sep;14(9):5223-35. doi: 10.1523/JNEUROSCI.14-09-05223.1994. PMID 8083732
- [Background] Spurrier J, Nicholson L, Fang XT, Stoner AJ, Toyonaga T, Holden D, Siegert TR, Laird W, Allnutt MA, Chiasseu M, Brody AH, Takahashi H, Nies SH, Perez-Canamas A, Sadasivam P, Lee S, Li S, Zhang L, Huang YH, Carson RE, Cai Z, Strittmatter SM. Reversal of synapse loss in Alzheimer mouse models by targeting mGluR5 to prevent synaptic tagging by C1Q. Sci Transl Med. 2022 Jun;14(647):eabi8593. doi: 10.1126/scitranslmed.abi8593. Epub 2022 Jun 1. PMID 35648810
- [Background] Nabulsi NB, Mercier J, Holden D, Carre S, Najafzadeh S, Vandergeten MC, Lin SF, Deo A, Price N, Wood M, Lara-Jaime T, Montel F, Laruelle M, Carson RE, Hannestad J, Huang Y. Synthesis and Preclinical Evaluation of 11C-UCB-J as a PET Tracer for Imaging the Synaptic Vesicle Glycoprotein 2A in the Brain. J Nucl Med. 2016 May;57(5):777-84. doi: 10.2967/jnumed.115.168179. Epub 2016 Feb 4. PMID 26848175
- [Background] Naganawa M, Li S, Nabulsi N, Henry S, Zheng MQ, Pracitto R, Cai Z, Gao H, Kapinos M, Labaree D, Matuskey D, Huang Y, Carson RE. First-in-Human Evaluation of 18F-SynVesT-1, a Radioligand for PET Imaging of Synaptic Vesicle Glycoprotein 2A. J Nucl Med. 2021 Apr;62(4):561-567. doi: 10.2967/jnumed.120.249144. Epub 2020 Aug 28. PMID 32859701
- [Background] Li S, Cai Z, Wu X, Holden D, Pracitto R, Kapinos M, Gao H, Labaree D, Nabulsi N, Carson RE, Huang Y. Synthesis and in Vivo Evaluation of a Novel PET Radiotracer for Imaging of Synaptic Vesicle Glycoprotein 2A (SV2A) in Nonhuman Primates. ACS Chem Neurosci. 2019 Mar 20;10(3):1544-1554. doi: 10.1021/acschemneuro.8b00526. Epub 2018 Nov 16. PMID 30396272
- [Background] Chen MK, Mecca AP, Naganawa M, Finnema SJ, Toyonaga T, Lin SF, Najafzadeh S, Ropchan J, Lu Y, McDonald JW, Michalak HR, Nabulsi NB, Arnsten AFT, Huang Y, Carson RE, van Dyck CH. Assessing Synaptic Density in Alzheimer Disease With Synaptic Vesicle Glycoprotein 2A Positron Emission Tomographic Imaging. JAMA Neurol. 2018 Oct 1;75(10):1215-1224. doi: 10.1001/jamaneurol.2018.1836. PMID 30014145